CLINICAL TRIAL: NCT03267355
Title: Indications and Outcomes of Gastrointestinal Endoscopic Ultrasound in Tanta-Egypt: Initial Experience.
Brief Title: Indications and Outcomes of Endoscopic Ultrasound in Tanta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EUS TANTA
Record Dates: First submitted 2017-08-27; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Gastric Disease; Intestinal Disease; Pancreatic Diseases; Esophageal Diseases
MeSH Terms: conditions — Stomach Diseases; Intestinal Diseases; Pancreatic Diseases; Esophageal Diseases | interventions — Endosonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastrointestinal diseases (Experimental): Endoscopic Ultrasound
  Interventions: Device: Endoscopic Ultrasound

INTERVENTIONS:
Device: Endoscopic Ultrasound — Indication of EUS
  Other Names: EUS

SUMMARY:
The aim is to evaluate the initial experience for the indications and outcomes of EUS in Tanta university hospital.

DETAILED DESCRIPTION:
Detection of main causes for referral to EUS in Tanta, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* All cases of gastrointestinal EUS

Exclusion Criteria:

* Missed data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of different indications for Endoscopic Ultrasound in Tanta, Egypt | 10 months
  Evaluation of the initial experience of the indications and outcomes of GIT EUS

CONTACTS AND LOCATIONS:
Overall Officials: Asem Elfert, Professor, Principal Investigator — Tanta University Faculty of Medicine; Ferial El-kalla, Professor, Principal Investigator — Tanta university Faculty of Medicine; Samah Mosaad, consultant, Study Director — Tanta University Faculty of Medicine; Walaa Elkhalawany, Consultant, Study Director — Tanta University Faculty of Medicine; Reham Elkhouly, Consultant, Study Chair — Tanta University Faculty of Medicine; Eslam Saber, Specialist, Study Chair — Tanta University Faculty of medicine
Locations (1):
- Tanta university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided